CLINICAL TRIAL: NCT00161408
Title: Psychological Intervention for Relapse Prevention in First Episode Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01GI9932-P2223
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenic Disorders
Keywords: schizophrenia, first episode, cognitive behavioural therapy, psychoeducation
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: cognitive behavioural therapy
Behavioral: psychoeducation

SUMMARY:
The study is a randomized clinical trial investigating the efficacy of a comprehensive psychological intervention for the treatment of first episode schizophrenia

DETAILED DESCRIPTION:
Patients suffering from their first episode of schizophrenic disorders are randomly allocated to either a short "information centered psychoeducation" (ICP) of 8 sessions or a "cognitive behavioral treatment" (CBT). CBT includes 8 sessions of psychoeducation, 8 sessions of computer based cognitive training, 8 sessions with relatives and 20 sessions of focusing on stress management, relapse prevention and coping with persistent symptoms.

The primary endpoint is relapse at the one and two year follow up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenic disorder according to ICD 10: F20
* first episode
* age between 18 and 55
* willingness to give informed consent also to a double blind pharmacological treatment study

Exclusion Criteria:

* residence outside of the catchment area
* insufficient knowledge of the German language
* substance abuse or addiction as primary clinical problem
* serious physical illness
* organic brain disease
* pregnancy
* contraindications to neuroleptic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106
Dates: Start 2000-12; Study Completion 2005-09

PRIMARY OUTCOMES:
relapse

SECONDARY OUTCOMES:
quantitative measures of symptoms
social functioning
cognitive functioning
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klingberg, PD Dr. phil. Dipl. Psych., Principal Investigator — University Hospital Tuebingen
Locations (5):
- Germany (5):
  - Department of Psychiatry and Psychotherapy, University of Bonn, Bonn
  - Department of Psychiatry and Psychotherapy, University of Cologne, Cologne
  - Department of Psychiatry and Psychotherapy, University of Duesseldorf, Düsseldorf
  - Department of Psychiatry and Psychotheray, University of Muenchen, München
  - Department of Psychiatry and Psychotherapy, University of Tuebingen, Tübingen